CLINICAL TRIAL: NCT07257718
Title: The Combined Role of FAPI PET and Liquid Biopsy in the Staging and Clinical Management of Bladder Cancer
Brief Title: The Combined Role of FAPI PET and Liquid Biopsy in the Staging and Clinical Management of Bladder Cancer - FUTURE Trial
Acronym: FUTURE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chiti Arturo (Other)
Responsible Party: Sponsor-Investigator, Chiti Arturo, Professor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FUTURE
Record Dates: First submitted 2025-11-18; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Liquid Biopsy; Cystectomy; Conservative Treatment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BC patients eligible for radical cystectomy (Experimental): BC patients treated with radical cystectomy ± neoadjuvant therapy
  Interventions: Procedure: FAPI PET/CT and liquid biopsy in patients eligible for radical cystectomy
- BC patients treated with systemic therapy (Experimental): patients eligible for conservative treatment
  Interventions: Procedure: FAPI PET/CT and liquid biopsy in patients eligible for conservative treatment

INTERVENTIONS:
Procedure: FAPI PET/CT and liquid biopsy in patients eligible for radical cystectomy — We hypothesise that FAPI PET improves clinical staging, and that baseline FAPI PET metrics and ctDNA/utDNA profiles correlate with tumour aggressiveness and patient outcomes
  Arms: BC patients eligible for radical cystectomy
Procedure: FAPI PET/CT and liquid biopsy in patients eligible for conservative treatment — We hypothesise that FAPI PET improves clinical staging, and that baseline FAPI PET metrics and ctDNA/utDNA profiles correlate with tumour aggressiveness and patient outcomes
  Arms: BC patients treated with systemic therapy

SUMMARY:
The study will be a prospective two arms diagnostic phase II single-center trial.

Patients referred for diagnosis and treatment with diagnosis of bladder cancer, age > 18 years, ECOG performance status < 2, ability to undergo an imaging study procedure will be considered for inclusion. For the study will be include 262 patients (118 and 144 in the arm 1 and 2, respectively).

Eligible patients will sign the inform consent to be included in the study. The participation to other clinical studies will be not, per se, an exclusion criterion. Before treatment, enrolled patients will be imaged by FAPI PET/CT and urine samples will be collected and analyzed by Epicheck® test and Xpert® Bladder Cancer Detection. Thereafter, patients will be managed and treated according to international guidelines and standard of care procedures in our institution. Safety will be recorded. Results of FAPI imaging, Epicheck® test, and Xpert® Bladder Cancer Detection will be compared to stage, risk assessment groups as defined by currentguidelines, and clinical outcome. Diagnostic and predictive performances of FAPI imaging and liquid biopsy will be assessed and compared by using machine learning approaches.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* ECOG performance status < 2
* ability to undergo an imaging study procedure

Exclusion Criteria:

* pregnant or breast-feeding women
* uncontrolled active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of FAPI PET/CT for the detection in the Staging of Bladder Cancer | from enrollment to 48 months
  Sensitivity will be calculated as the proportion of true positive findings obtained with FAPI PET/CT compared with the reference standard (e.g., clinical follow-up).

SECONDARY OUTCOMES:
PET Imaging | from month 12 to 60
  secondary outcome aims to image patients

CONTACTS AND LOCATIONS:
Overall Officials: Martina Sollini, Principal Investigator — IRCCS Ospedale San Raffaele

IPD SHARING:
Plan to Share IPD: Undecided